CLINICAL TRIAL: NCT01035164
Title: Open-label, Non-randomized, Positron Emission Tomography (PET) Imaging Study to Evaluate a Single Dose of 250 MBq (6.75 mCi) ZK 6032924 (18F-FEDAA1106) for Its Diagnostic Potential in Discriminating Patients With Probable Alzheimer's Disease From Healthy Volunteers and to Evaluate the Radiation Dosimetry of a Single Dose of 185 MBq (5 mCi) ZK 6032924 in Healthy Volunteers.
Brief Title: Evaluation of ZK 6032924 in Probable Alzheimer's Disease Patients Versus Healthy Volunteers and the Radiation Dosimetry of ZK 6032924 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91683; 2006-006045-14 (EudraCT Number); 311401
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Positron-Emission Tomography; Alzheimer's Disease
Keywords: Alzheimer's Disease; Diagnostic Imaging; Neuroinflammation; PET Diagnosis; PET Tracer
MeSH Terms: conditions — Alzheimer Disease; Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: F-18 FEDAA1106 (BAY85-8101)
- Arm 2 (Experimental)
  Interventions: Drug: F-18 FEDAA1106 (BAY85-8101)
- Arm 3 (Experimental)
  Interventions: Drug: F-18 FEDAA1106 (BAY85-8101)

INTERVENTIONS:
Drug: F-18 FEDAA1106 (BAY85-8101) — Alzheimer Disease patients: Single intravenous bolus injection of 250 MBq BAY85-8101 on day one of the treatment period, PET
  Arms: Arm 1
Drug: F-18 FEDAA1106 (BAY85-8101) — Healthy volunteers for brain imaging: Single intravenous bolus injection of 250 MBq BAY85-8101 on day one of the treatment period, PET
  Arms: Arm 2
Drug: F-18 FEDAA1106 (BAY85-8101) — Healthy volunteers for whole body imaging: Single intravenous bolus injection of 185 MBq BAY85-8101, whole body PET for evaluation of effective dose, kinetics of BAY85-8101 in blood
  Arms: Arm 3

SUMMARY:
PET (positron emission tomography) imaging with BAY85-8101 (ZK 6032924) in patients with Alzheimer's Disease compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:Patients for brain imaging:- patient and designee capable of giving fully informed consent in writing- patient fulfils DSM-IV and NINCDS-ADRDA criteria for probable Alzheimer's disease. Other forms of dementia excluded- males or postmenopausal females aged >/= 50 yearsHealthy volunteers for brain imaging: - able to give fully informed consent in writing- absence of any sign of dementia/cognitive impairment in neuropsychological examinations- males or postmenopausal females aged >/= 50 years Healthy volunteers for whole body imaging:- able to give fully informed consent in writing - males or postmenopausal females aged >/= 60 years - no significant disease or drug use Exclusion Criteria:For all healthy volunteers and patients:- Any disease, condition, or concomitant medications that significantly compromises the function of the body systems and could result in excessive accumulation, impaired metabolism, altered excretion of the radiotracer, or might interfere with the conduct of the study or interpretation of the results

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Visual analysis/description of the uptake and description of brain PET scans | Day of study tracer administration
Standardized uptake value (SUV) in various cerebral regions/volumes of interest (ROI/VOI) assumed and found to be involved in the pathophysiology of Alzheimer's disease. | Day of study tracer administration

SECONDARY OUTCOMES:
Standard quantification variables derived from 3D PET imaging and brain modeling | Day of study tracer administration
Standard Safety Measurement:adverse event collection | Maximum time from Screening to Follow up are 37 days
Standard Safety Measurement:electrocardiogram | Maximum time from Screening to Follow up are 37 days
Standard Safety Measurement:safety laboratory | Maximum time from Screening to Follow up are 37 days
Standard Safety Measurement: vital signs | Maximum time from Screening to Follow up are 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Amsterdam, Netherlands
- Stockholm, Sweden

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/